CLINICAL TRIAL: NCT04157322
Title: 5-hydroxymethylation Signatures in Plasma Circulating Cell-free DNA as Markers for Tumor Burden and Recurrence in Appendiceal and Colorectal Peritoneal Metastasis
Brief Title: Plasma 5hmC Signatures as a Marker of Colorectal / Appendiceal Peritoneal Metastasis
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB19-0913
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer Stage IV; Colorectal Cancer Metastatic; Colorectal Cancer, Genetics of; Appendix Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Appendiceal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: prospective single arm biomarker (plasma cell-free DNA hydroxymethylation) study — Blood draw

SUMMARY:
Patients with peritoneal metastasis of colorectal or high grade appendiceal origin who are candidates for cytoreductive surgery with HIPEC (hyperthermic intraperitoneal chemotherapy) will be enrolled in this study. Blood collection for measurements of plasma cell-free DNA hydroxymethylation signatures will be performed at different time points, before and after surgery, in order to determine if plasma hydroxymethylation signatures are more sensitive than conventional tumor markers in identifying clinically detectable recurrence at 1 year after surgery.

DETAILED DESCRIPTION:
This will be a prospective single arm biomarker (plasma-free DNA 5-hydroxymethylation) study. Fifty-five Adult patients with peritoneal metastases of colorectal and appendiceal origin who are candidates for a curative surgery and fulfill the inclusion criteria will be offered to participate in this study. In addition to the postoperative standard of care oncological surveillance of these patients which includes periodic physical examinations, cross sectional imaging studies (CT or MRI) and blood work for conventional tumor markers, serial measurements of plasma hydroxymethylation signatures will be performed. We will use a model developed in a separate pilot study to identify recurrent peritoneal metastasis based on 5hmC signatures. As part of this study, blood collection for measurements of plasma hydroxymethylation signatures of target genes will be performed at seven time points:

* Just before surgery (During the preoperative clinic visit or at the operating room).
* 5-7 days after surgery (just before hospital discharge).
* 6 weeks after surgery (first postoperative clinic visit).
* 3 months after surgery (second postoperative clinic visit).
* 6 months after surgery (third postoperative clinic visit).
* 9 months after surgery (fourth postoperative clinic visit).
* 12 months after surgery (fifth postoperative clinic visit). Standard of care surveillance elements that include patient history and physical examination, conventional blood biomarkers (CEA, CA 19-9 and CA 125) and cross sectional imaging of the chest, abdomen and pelvis will be undertaken simultaneously at similar time points. We will then compare the sensitivities of DNA hydroxymethylation signatures and conventional blood biomarkers in diagnosing clinically detectable recurrence at 1 year after surgery. We hypothesize that plasma hydroxymethylation signatures have higher sensitivity in identifying clinically detectable recurrence when compared with conventional tumor markers (CEA, CA 19-9 and CA 125).

ELIGIBILITY:
Inclusion Criteria:

I. Histologic proof of colorectal adenocarcinoma or high grade appendiceal tumors (appendiceal adenocarcinoma or ex-goblet adenocarcinoma Tang B or C).

II. Age ≥ 18 years. III. Patients with known peritoneal metastasis (PM) who are candidates for complete cytoreduction and HIPEC. Known PM - diagnosed previously by diagnostic laparoscopy / laparotomy or clear radiological evidence of PM.

IV. Neoadjuvant chemotherapy permitted. V. The patient is able to provide informed consent. VI. The patient is planned to undergo his / her postoperative surveillance at UCM, as this study's protocol requires multiple clinic visits.

VII. No evidence of systemic metastasis.

-

Exclusion Criteria:

Vulnerable subjects will not participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with peritoneal metastasis of colorectal or high grade appendiceal origin who are candidates for cytoreductive surgery with hyperthermic intraperitoneal chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
clinically detectable recurrence at 1 year after surgery. | 5 years
  1. Clear radiological evidence of recurrent disease.
  2. Histopathological proof (by means of endoscopy, imaging guided biopsy or diagnostic surgery) of recurrent disease.
  3. A new lesion revealed by physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Bissonnette, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided